CLINICAL TRIAL: NCT01904825
Title: Use of Sentinel Cells for the Development of Molecular Tests to Control the Quality of Cryopreservation
Status: Withdrawn | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: Bonnin PHRC IR 2006
Record Dates: First submitted 2013-07-12; First posted 2013-07-22 (Estimated); Last update posted 2013-07-22 (Estimated); Status verified 2013-07

CONDITIONS: Aneurysm of the Abdominal Aorta

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day

SUMMARY:
The aim is to set up tools that will serve as quality tracers for cryopreservation procedures.

To meet this objective, we have chosen to develop reference samples (sentinel cells) that, in the medium term, can be used as controls to guarantee the quality of preservation for biological samples.

The biological tools and an optimised follow-up strategy will make it possible to validate preservation procedures at the CRB in order to guarantee the perfect stability of samples and the validity of clinical studies.

ELIGIBILITY:
Inclusion Criteria:

* Age > or = 18 years
* All patients presenting an abdominal aorta diameter of at least 5 cm at the time of discovery and who have surgery

Exclusion Criteria:

* Patients who do not have aneurysm of the abdominal aorta
* Refusal to sign the consent form for participation
* Patients who do not wish to have their operation in Dijon or Strasbourg CHU

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Only patients of the CHU Dijon and Strasbourg
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2006-09; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Quality sentinel cells | participants will be followed for the duration of hospital stay, an expected average of 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Alain BONNIN, Principal Investigator — CHU Dijon - Biological Resource Center